CLINICAL TRIAL: NCT06613373
Title: An Exploratory Clinical Study of CDK4/6i Dalpiciclib Combined With AI Neoadjuvant Therapy for Stage II-III HR+/HER2- Breast Cancer
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Jiangsu Famous Medical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OBU-BC-II-093
Record Dates: First submitted 2024-09-20; First posted 2024-09-25 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — dalpiciclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experimental (Experimental): Dalpiciclib combined with AI,28 days as one cycle.
  Dalpiciclib: 150 mg (p.o.) was given once daily for 3 weeks, followed by 1 week off in each 4-week cycle.
  Letrozole: 2.5mg, p.o., once a day, continuous administration.
  Interventions: Drug: Dalpiciclib

INTERVENTIONS:
Drug: Dalpiciclib — Dalpiciclib: 150 mg (p.o.) was given once daily for 3 weeks, followed by 1 week off in each 4-week cycle.

SUMMARY:
This is a single-arm, open-label, exploratory clinical study

DETAILED DESCRIPTION:
This is a single-arm, open-label, exploratory clinical study initiated by the investigator to evaluate the objective response rate (ORR), efficacy, and safety of Dalpiciclib combined with AI in the neoadjuvant treatment of stage Ⅱ-Ⅲ HR+/HER2- breast cancer.

ELIGIBILITY:
Inclusion Criteria:

-

1. For premenopausal or postmenopausal women, the definition of menopause:

1. previous bilateral oophorectomy, or age ≥60 years; or
2. Age <60, natural postmenopausal status (defined as spontaneous cessation of regular menstruation for at least 12 consecutive months without other pathological or physiological causes), E2 and FSH at postmenopausal levels; 2. All patients had estrogen receptor (ER) positive (> 10%), HER2 receptor-negative invasive breast cancer regardless of PR expression level. Follow the 2018 ASC-CAP HER2 Negative Interpretation Guidelines. Immunohistochemical (IHC) scores of 0+ or 2+ and in situ hybridization (ISH) test negative were confirmed by pathology laboratory (HER-2/CEP17 ratio < 2.0); 3. Patients with initial treatment of stage II-III whose tumor stage meets AJCC 8th edition standard; 4. There is no known severe hypersensitivity to compounds or endocrine therapy similar to Darcilil or darcilil excipients.

5. ECOG 0-1; 6. The patient must be able to swallow oral medications. 7. The functional level of the organ must meet the following requirements:

1. Bone marrow function ANC ≥ 1.5×109/L (no growth factor used within 14 days); PLT ≥ 100×109/L (no corrective therapy used within 7 days); Hb ≥ 100 g/L (no corrective therapy used within 7 days);
2. Liver and kidney function TBIL≤1.5×ULN; ALT and AST≤3×ULN (ALT and AST≤5×ULN in patients with liver metastasis); BUN and Cr≤1.5×ULN and creatinine clearance ≥50 mL/min (Cockcroft-Gault formula);
3. 12-lead electrocardiogram QT interval ≤480 ms; 8. Able to accept all needle biopsies required by the protocol; 9. Voluntarily participate in this study, sign informed consent, have good compliance and be willing to cooperate with follow-up.

Exclusion Criteria:

1. Previously received any form of anti-tumor therapy (chemotherapy, radiotherapy, molecular targeted therapy, endocrine therapy, etc.);
2. At the same time receive any anti-tumor treatment other than that prescribed in other protocols;
3. Bilateral breast cancer, inflammatory breast cancer or ocessive breast cancer;
4. Stage IV breast cancer;
5. Other malignant tumors have appeared in the past 5 years;
6. Severe heart, liver, kidney and other vital organ dysfunction;
7. Inability to swallow, chronic diarrhea, and intestinal obstruction, with multiple factors affecting drug use and absorption;
8. Known allergic history of the drug components of this protocol; Have a history of immunodeficiency, including HIV positive, HCV, active viral hepatitis B or other acquired, congenital immunodeficiency diseases, or a history of organ transplantation;
9. Pregnant and lactating women, fertile women who tested positive for baseline pregnancy tests, or women of childbearing age who were unwilling to take effective contraceptive measures during the entire test period;
10. Concomitant diseases (including but not limited to severe high blood pressure, severe diabetes, active infection, etc.) that, in the judgment of the investigator, seriously endanger the patient's safety or affect the patient's ability to complete the study;
11. Have a clear history of neurological or mental disorders, including epilepsy or dementia. The investigator did not consider the patient suitable for participation in any other condition of the study.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-10-15 (Estimated); Primary Completion 2025-10-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
ORR | 24 month
  Objective response rate

IPD SHARING:
Plan to Share IPD: No